CLINICAL TRIAL: NCT02192541
Title: Phase I Study of Ganetespib and Ziv-Aflibercept in Patients With Advanced Gastrointestinal Carcinomas, Non-Squamous Non-Small Cell Lung Carcinomas, Urothelial Carcinomas, and Sarcomas
Brief Title: Ganetespib and Ziv-Aflibercept in Refractory Gastrointestinal Carcinomas, Non-Squamous Non-Small Cell Lung Carcinomas, Urothelial Carcinomas, and Sarcomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supplier suspended further clinical development of Ganetespib
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140150; 14-C-0150
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Neoplasms
Keywords: Urothelial Carcinomas; Non-Squamous Non-Small Cell Lung Carcinomas; Refractory Gastrointestinal Carcinomas; Hsp90 Inhibitor; Sarcomas
MeSH Terms: conditions — Neoplasms; Sarcoma | interventions — aflibercept; STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ganetespib and Ziv-Aflibercept (Experimental): Ganetespib was administered intravenously, over 1 hour, weekly, on days 1, 8, and 15 of each 28-day cycle. Ziv-aflibercept was administered intravenously, over 1 hour, every 2 weeks, on days 1 and 15 of each 28-day cycle. Ganetespib was started at a dose level of 100 mg/m^2 + ziv-aflibercept at 3 mg/kg or 4 mg/kg.
  Interventions: Drug: Ziv-Aflibercept; Drug: Ganetespib

INTERVENTIONS:
Drug: Ziv-Aflibercept — Ziv-aflibercept is a soluble fusion protein with high binding affinity for vascular endothelial growth factor A (VEGF-A), vascular endothelial growth factor B (VEGF-B), and placenta growth factor (PIGF) and thus confers anti-angiogenic activity
  Other Names: ZALTRAP; VEGF-TRAP
Drug: Ganetespib — Ganetespib is a non-geldamycin synthetic inhibitor of Hsp90 with activity against multiple cancer cell lines and tumor xenografts in preclinical models.
  Other Names: STA-9090

SUMMARY:
Background:

- Some people have cancers that don't respond to standard treatments. In these cases, doctors may try to use drugs to slow the growth of the cancer.

Objectives:

- To test the safety and efficacy of the drug combination of ganetespib and ziv-aflibercept.

Eligibility:

- Adults age 18 and over with advanced cancer of the colon, lung, urinary tract, and sarcomas.

Design:

* Participants will be screened with medical history, blood tests, and scans to measure their tumors.
* Participants will have one or two eye exams, with dilating eye drops.
* Participants will get the study drugs at the clinic as an infusion in a vein. Ganetespib will be given once a week on the same day for 3 weeks in a row, followed by a 1-week rest period. Ziv-aflibercept will be given once every other week. The drugs will be given in 28-day cycles.
* Participants may have a small piece of their tumor collected once or twice. This is done using a small needle during computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound scan.
* Participants will have their blood pressure checked at each visit. They will check it at home every day of the study.
* Participants may have one or more whole-body positron emission tomography (PET) scans with 89Zr-panitumumab. A small amount of a radioactive chemical will be injected through a tube in an arm. Participants will lie on a bed that slides in and out of the donut-shaped PET scanner. They will have small amounts of blood drawn.
* Participants may stay in the study as long as they are tolerating the drugs and their tumor is not getting worse.

DETAILED DESCRIPTION:
BACKGROUND:

* Ganetespib is a non-geldamycin synthetic inhibitor of Hsp90 that has demonstrated activity against multiple cancer cell lines and tumor xenografts in preclinical models. Inhibiting the Hsp90 chaperone complex results in the recruitment of ubiquitin ligases, polyubiquination, and proteosomal degradation of Hsp90 client proteins, including transcription factors and proteins involved in angiogenesis vascular endothelial growth factor (VEGF), vascular endothelial growth factor receptor (VEGFR), hypoxia-inducible factor 1 (HIF-1), signal transducers and activators of transcription protein 3 (STAT-3); growth factor independence rapidly accelerated fibrosarcoma (RAF), epidermal growth factor receptor (EGFR), human epidermal growth factor receptor 2 (Her2), insulin-like growth factor 1 receptor (IGFR); resistance to anti-growth signals cyclin-dependent kinase 4 (CDK4); tissue invasion and metastases mesenchymal-epithelial transition factor (MET), matrix metalloproteinase-2 (MMP2); and avoidance of apoptosis protein kinase B (AKT), rat insulin promoter (RIP), Survivin, B cell lymphoma (Bcl-2).
* HIF-1-alpha activation has been implicated in mediating resistance to anti-angiogenic therapy; recent evidence implicates a greater role for Hsp90 in direct modulation of VEGF signaling.
* Combining Hsp90 inhibition with ganetespib and anti-angiogenic therapy with Ziv-Aflibercept, a soluble fusion protein with high binding affinity for vascular endothelial growth factor A (VEGF-A), vascular endothelial growth factor B (VEGF-B), and placenta growth factor (PIGF), presents a rational novel strategy for improving upon and overcoming resistance to anti-angiogenic therapy

PRIMARY OBJECTIVE:

- To establish the safety, tolerability, and maximum tolerated dose (MTD) of the combination of ganetespib and Ziv-Aflibercept in patients with refractory gastrointestinal carcinomas, non-squamous non-small cell lung carcinomas, urothelial carcinomas, and sarcomas

SECONDARY OBJECTIVE:

* To assess modulation of HIF-1-alpha as a pharmacodynamic marker of therapy with the combination of ganetespib and Ziv-Aflibercept
* To assess modulation of epidermal growth factor receptor (EGFR) expression using 89Zr-labeled, EGFR-targeting antibody panitumumab positron emission tomography (PET)/computed tomography (CT) imaging of tumor lesions prior to and following treatment with study drugs

ELIGIBILITY:

* Adult patients with histologically confirmed metastatic gastrointestinal carcinomas, non-squamous non-small cell lung carcinomas, urothelial carcinomas, and sarcomas with disease progression after at least one line of standard therapy
* Participants in the expansion phase must demonstrate EGFR expression on archival tumor samples and have disease amenable to biopsy with willingness to undergo pre- and post-treatment biopsies
* No major surgery within 4 weeks prior to study enrollment, no radiation or chemotherapy within 3 weeks prior to enrollment; patients must have recovered from toxicities of prior therapies to at least eligibility levels prior to enrollment.

STUDY DESIGN:

* Ganetespib will be administered intravenously weekly on days 1, 8, and 15 of a 28-day cycle. Ziv-Aflibercept will be administered intravenously every 2 weeks, on days 1 and 15, during a 28-day cycle.
* The escalation portion of the trial will follow a standard 3+3 design, whereby patients are dose-escalated in cohorts of 3 until dose-limiting toxicity is observed.
* Once the MTD is established, 10 additional patients will be enrolled to the expansion phase, at the MTD, and tumor biopsies will be obtained to assess pharmacodynamic endpoints. During cycle 1 of the expansion phase, ganetespib will be administered intravenously weekly, on days 8 and 15 with omission of day 1 treatment to accommodate a baseline biopsy pre-ganetespib but after administration of Ziv-Aflibercept. For all subsequent cycles, ganetespib will be administered days 1, 8, and 15. Ziv-Aflibercept will still be administered intravenously every 2 weeks, on days 1 and 15, of a 28-day cycle.
* PET/CT imaging with 89Zr-labeled panitumumab will be performed to evaluate tumor distribution prior to and following treatment with study agents.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histologically confirmed recurrent or metastatic gastrointestinal carcinomas, non-squamous non-small cell lung carcinomas, urothelial carcinomas, and sarcomas with disease progression after at least one line of standard therapy. Disease should have progressed following all treatments known to prolong survival, unless a given treatment is contraindicated.

* Patients with colorectal carcinoma must have progressed through at least two lines of standard chemotherapy in the metastatic setting.
* Patients with non-small cell lung cancer with known sensitizing epidermal growth factor receptor (EGFR) mutation and/or anaplastic lymphoma receptor tyrosine kinase (ALK) rearrangement should have received prior erlotinib and/or crizotinib, respectively.
* Patients with urothelial carcinoma will have progressed on prior platinum-based therapy or for which platinum-based therapy is contraindicated.
* Patients enrolled on the expansion phase of the protocol must demonstrate EGFR expression by immunohistochemistry on archival tumor samples prior to undergoing (89) Zr-panitumumab positron emission tomography (PET)/computed tomography (CT) scans.

Age greater than or equal to 18 years of age.

Eastern Cooperative Oncology Group (ECOG) performance status < 2.

Life expectancy > 3 months.

Patients must have normal organ and marrow function as defined below:

* absolute neutrophil count greater than or equal to 1,500/mcL
* platelets greater than or equal to 100,000/mcL
* total bilirubin less than or equal to 1.5 times institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase SGOT)/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase SGPT) less than or equal to 3 times institutional upper limit of normal
* creatinine less than or equal to 1.2 times institutional upper limit of normal

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* urine protein/creatinine < 1 mg/mg
* International Normalized Ratio (INR) < 1.5

Cardiac function within institutional normal limits on echocardiogram.

Patients must have blood pressure no greater than 140 mmHg (systolic blood pressure) and 90 mmHg (diastolic blood pressure) for eligibility. Initiation or adjustment of antihypertensive medications is permitted prior to study entry provided that the average of three blood pressure measurements at enrollment visit is less than 140/90 mmHg.

The effects of ganetespib on the developing human fetus are unknown. For this reason and because anti-angiogenic agents similar to ziv-aflibercept are known to be teratogenic, women of child-bearing potential and men must agree to use two forms of contraception (hormonal or barrier method of birth control; abstinence; sterilization) prior to study entry, for the duration of study participation, and for 3 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use two forms of contraception prior to the study, for the duration of study participation, and for 3 months after completion of administration of both ganetespib and ziv-aflibercept.

Ability to understand and the willingness to sign a written informed consent document.

During the escalation phase of the protocol, patients may have evaluable or measurable disease. During the expansion phase of the protocol, patients must have 1) measurable disease, 2) disease amenable to biopsy and 3) willingness to undergo pre- and post-treatment biopsies.

EXCLUSION CRITERIA:

Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.

Patients who are receiving any other investigational agents.

Patients with known active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients whose brain metastatic disease status has remained stable for greater than or equal to 4 weeks following treatment of brain metastases are eligible to participate at the discretion of the principal investigator.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active untreated infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Patients with known serious cardiac illness or medical conditions, including but not

limited to:

* Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, unstable angina or history of myocardial infarct within 6 months prior to enrollment, or indwelling temporary pacemaker
* Ventricular tachycardia or a supraventricular tachycardia that requires treatment with antiarrhythmic agents
* Second- or third-degree atrioventricular block unless treated with a permanent pacemaker
* Complete left bundle branch block
* History of long Q wave, T wave (QT) syndrome or a family member with this condition

No major surgery within 4 weeks prior to enrollment or history of gastrointestinal bleeding within 3 months prior to enrollment. No signs or symptoms of active bleeding or nonhealing ulcer will be permitted at study entry. Patients with central pulmonary tumors with evidence of bronchial invasion, or presenting with hemoptysis will be excluded.

Corrected QT interval (QTc) > 470 msec on electrocardiogram (by Bazett's; average of triplicate recordings at the discretion of the principal investigator (PI) will exclude patients from entry on study. Medications that are known to cause QTc interval prolongation are prohibited for patients entering on trial. Patients for whom a given medication that may cause QTc interval prolongation cannot be discontinued, may be eligible at the discretion of the study PI, provided QTc interval criteria is met at enrollment. A comprehensive list of agents with the potential to cause QTc prolongation can be found in Appendix C and at http://crediblemeds.org.

Pregnant women and women who are breastfeeding are excluded from this study because the effects of the study drugs on the developing fetus are unknown.

Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ganetespib and zivaflibercept. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Substrates of cytochrome P450 3A4 (CYP3A4) or cytochrome P450 2C19 (CYP2C19):

* Preliminary results of a clinical drug-drug interaction study, examining the effect of ganetespib on the pharmacokinetics of the CYP2C19-sensitive probe omeprazole, show a modest (20%) increase in omeprazole exposure when coadministered with ganetespib.
* In vitro data implies expectation of greater interaction with CYP2C19 substrates than with CYP3A4 substrates.
* Caution is advised when sensitive narrow therapeutic range CYP3A4 or CYP2C19 substrates are concomitantly administered.

Inhibitors of P-Glycoprotein Efflux Transporters: Concomitant medications that are strong inhibitors of P-glycoprotein efflux transporters should be used with caution during the study; examples of these medications include:

* ritonavir,
* cyclosporine,
* verapamil,
* erythromycin,
* ketoconazole,
* itraconazole,
* quinidine, and
* elacridar.

Concurrent anticoagulation will be permitted providing the patient is receiving a stable dose of anticoagulants before study entry. Patients receiving anticoagulants will be eligible for this trial. Evidence of clinically significant bleeding diathesis or underlying coagulopathy (e.g., INR > 1.5 without vitamin K antagonist therapy) will not be permitted.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Bottsford-Miller JN, Coleman RL, Sood AK. Resistance and escape from antiangiogenesis therapy: clinical implications and future strategies. J Clin Oncol. 2012 Nov 10;30(32):4026-34. doi: 10.1200/JCO.2012.41.9242. Epub 2012 Sep 24. PMID 23008289
- [Background] Stravopodis DJ, Margaritis LH, Voutsinas GE. Drug-mediated targeted disruption of multiple protein activities through functional inhibition of the Hsp90 chaperone complex. Curr Med Chem. 2007;14(29):3122-38. doi: 10.2174/092986707782793925. PMID 18220746
- [Derived] Meehan R, Kummar S, Do K, O'Sullivan Coyne G, Juwara L, Zlott J, Rubinstein L, Doroshow JH, Chen AP. A Phase I Study of Ganetespib and Ziv-Aflibercept in Patients with Advanced Carcinomas and Sarcomas. Oncologist. 2018 Nov;23(11):1269-e125. doi: 10.1634/theoncologist.2018-0203. Epub 2018 May 31. PMID 29853657
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0150.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The escalation of dose was not performed as planned for this study due to toxicity and early termination of the trial.
Groups:
- Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg: Ganetespib was administered intravenously, over 1 hour, weekly, on days 1, 8, and 15 of each 28-day cycle. Ziv-aflibercept was administered intravenously, over 1 hour, every 2 weeks, on days 1 and 15 of each 28-day cycle. Ganetespib was started at a dose level of 100 mg/m^2 and ziv-aflibercept at 4 mg/kg.
- Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg: Ganetespib was administered intravenously, over 1 hour, weekly, on days 1, 8, and 15 of each 28-day cycle. Ziv-aflibercept was administered intravenously, over 1 hour, every 2 weeks, on days 1 and 15 of each 28-day cycle. Ganetespib was administered at a level of 100 mg/m^2 and ziv-aflibercept at 3 mg/kg.
Period: Overall Study
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Started | 2 | 3
Treated | 2 | 3
Evaluable for Response | 1 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 59 [51 to 67] | 60 [50 to 63] | 60 [50 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
Diagnosis [Count of Participants; unit: Participants]
  Colon adenocarcinomas | 1 | 2 | 3
  Small bowel adenocarcinomas | 0 | 1 | 1
  Rectal adenocarcinomas | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status is graded on a scale of 0 to 5, with higher scores indicating lower levels of functioning in terms of ability to care for oneself, daily activities, and physical abilities (walking, working, etc.).
  Participants
    0: Fully active | 0 | 0 | 0
    1: Restricted in physically strenuous activity | 2 | 3 | 5
    2: Unable to carry out any work activities | 0 | 0 | 0
    3: Capable of only limited self-care | 0 | 0 | 0
    4: Completely disabled | 0 | 0 | 0
    5: Dead | 0 | 0 | 0
Number of Prior Therapies [Median (Full Range); unit: prior therapies] | 6.5 [5 to 8] | 8 [6 to 15] | 8 [5 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Regardless of Attribution Assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v4.0
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 12 months and 44 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

2. Primary Outcome: Number of Participants With Grade 2 or Greater Adverse Events Possibly, Probably, or Definitely Related to Administration of the Study Drugs
Description: Adverse Events were graded according to Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. Grade refers to the severity of the Adverse Event. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event (AE). AEs were considered possibly attributable to both study drugs, except where otherwise noted. Star (*) symbol indicates that the AE is possibly related to Ziv-aflibercept and unlikely to be related to Ganetespib.
Time Frame: Date treatment consent signed to date off study, approximately 12 months and 44 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 2 | 3
Participants
  Grade 2 Alanine Aminotransferase Increased | 0 | 1
  Grade 2 Anorexia | 1 | 0
  Grade 2 Diarrhea | 1 | 0
  Grade 2 EKG QT Corrected Interval Prolonged | 1 | 0
  Grade 2 Fatigue | 1 | 0
  Grade 2 Hypertension* | 0 | 1
  Grade 2 Hypocalcemia | 0 | 1
  Grade 2 Infusion Related Reaction | 1 | 0
  Grade 2 Lymphocycte Count Decreased | 0 | 1
  Grade 3 Abdominal Pain | 1 | 0
  Grade 3 Alkaline Phosphtase Increased | 0 | 1
  Grade 3 Gastritis* | 1 | 0
  Grade 5 Small Intestinal Perforation* | 1 | 0
  Grade 5 Sudden Death Not Otherwise Specified* | 0 | 1

3. Primary Outcome: Maximum Tolerated Dose (MTD) of the Combination of Ganetespib and Ziv-aflibercept
Description: MTD is defined as the dose level at which no more than 1 of 6 patients experience a dose limiting toxicity (DLT) during the first cycle of the treatment, and the dose level below that at which at least 2 (of <6) patients have a DLT as a result of the drug. Determination of DLT is based on the first cycle of treatment.
Time Frame: Cycle one (28 days)
Population: An MTD was not established because no MTD data were collected. The trial was terminated before the MTD was reached due to the decision of the drug supplier to suspend further clinical development of ganetespib.
Groups:
- Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg: Ganetespib was administered intravenously, over 1 hour, weekly, on days 1, 8, and 15 of each 28-day cycle. Ziv-aflibercept was administered intravenously, over 1 hour, every 2 weeks, on days 1 and 15 of each 28-day cycle. Ganetespib was started at a dose level of 100 mg/m^2 and ziv-aflibercept at 3 mg/kg.
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Modulation of Hypoxia-Inducible Factor 1 (HIF-1) Alpha
Description: To determine whether the combination of ganetespib and ziv-aflibercept modulated intratumoral Hypoxia-inducible factor 1 (HIF-1)-alpha expression, tumor biopsies were to be analyzed for change in HIF-1-alpha expression by immunofluorescence assay (IFA). Paired pre-and post-combination treatment samples were to be compared for qualitative changes in levels of HIF-1- alpha expression. Cores were to be normalized against the percentage of tumor within the sample.
Time Frame: Cycle 2, Day 7
Population: Data were not collected from any participant. Biopsies were to be collected from an expansion cohort treated at the maximum tolerated dose, after the conclusion of the dose escalation phase. Trial was closed before the MTD was established, patients were not enrolled to an expansion phase, and samples for pharmacodynamics analysis were not obtained.
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Modulation of Epidermal Growth Factor Receptor (EGFR) Expression
Description: To evaluate for tumor distribution of EGFR, patients were to undergo 89Zr-immuno-positron emission tomography (PET) imaging with 89Zr-labeled EGFR-targeting panitumumab antibody evaluate modulation of EGFR client protein prior to and after treatment with the combination of ganetespib and ziv-aflibercept. Panitumumab is a fully human monoclonal antibody that targets EGFR and competes with endogenous ligands to block stimulation of EGFR. 89z-immuno-PET imaging with panitumumab as a targeting ligand allows for quantification of EGFR within tumors.
Time Frame: Cycle 1 Day 16
Population: Data were not collected from any participant for this Outcome Measure. As the trial was closed before the maximum tolerated dose (MTD) was established, patients were not enrolled to an expansion phase, and samples for pharmacodynamics analysis were not obtained.
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants According to Best Response Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1)
Description: Radiologic response assessments by computed tomography (CT) scans were performed at baseline and every two cycles to evaluate tumor response based on the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria for target lesions: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progressive Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: Baseline and every 2 months up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 1 | 3
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 0 | 3
  Progressive Disease | 1 | 0

7. Secondary Outcome: Number of Cycles on Treatment
Description: The number of 28-day treatment cycles (ganetespib on days 1, 8, and 15; ziv-aflibercept on days 1 and 15) administered to each evaluable patient. Number represents treatment cycles that were started; not all cycles were completed.
Time Frame: up to 5 months
Population: The number of participants who were evaluable for response
Measure: Median (Full Range); unit: cycles
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 1 | 3
cycles | 1 [1 to 1] | 4 [4 to 5]

8. Other Pre Specified Outcome: Number of Participants Who Had a Dose Limiting Toxicity (DLT)
Description: A DLT is defined as an adverse event that is related (possibly, probably, or definitely) to administration of study drugs during cycle one and is a Grade ≥ 3 non-hematological toxicity. Grade ≥3 non-hematological toxicity felt to be related to study medications are: Grade 3 diarrhea if it is refractory to treatment; Grade 3 nausea and vomiting if it is refractory to anti-emetic therapy and unable to be corrected; rise in creatinine to Grade 3, not corrected to Grade 1 or less within 48 hours with intravenous (IV) fluids; Any Grade 4 corrected QT interval (QTc) prolongation; Grade 4 neutropenia ≥5 days or febrile neutropenia,...).
Time Frame: Cycle one (28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 12 months and 44 days
Arm/Group | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg (N=2) | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg (N=3)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 5, Stent placement; surgical complications (unlikely related to study drugs)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 5, possibly related to Ziv-Aflibercept
Sudden death Not Otherwise Specified (General disorders) | 0 (0) | 1 (1) — Grade 5, possibly related to Ziv-Aflibercept
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 4 mg/kg (N=2) | Dose Level -1: Ganetespib 100 mg/m^2 + Ziv-Aflibercept 3 mg/kg (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) — Grade 3, possibly related to study drugs
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1, possibly related to study drugs
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2, unlikely related to study drugs
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to Ziv-Aflibercept
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (2) — Grade 1, unlikely related to study drugs
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) — Grade 1, possibly related to study drugs
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) — Grade 2, possibly related to study drugs
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) — Grade 3, possibly related to study drugs
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) — Grade 2, unlikely related to study drugs
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to study drugs
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — Grade 1, possibly related to study drugs
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (3) — Grade 1, possibly related to study drugs
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — Grade 1, unlikely related to study drugs
Blurred vision (Eye disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2, unlikely related to study drugs
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Creatinine increased (Investigations) | 0 (0) | 2 (2) — Grade 1, possibly related to Ziv-Aflibercept
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2, unlikely related to study drugs
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (8) — Grade 1, possibly related to study drugs
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to study drugs
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to study drugs
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 1 (2) — Grade 1, possibly related to study drugs
Eye infection (Infections and infestations) | 0 (0) | 1 (1) — Grade 2, unlikely related to study drugs
Fatigue (General disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to study drugs
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3, possibly related to Ziv-Aflibercept
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) — Grade 1, possibly related to Ziv-Aflibercept
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 1, unlikely related to study drugs
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Hypertension (Vascular disorders) | 1 (1) | 1 (1) — Grade 2, unlikely related to study drugs
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — Grade 1, unlikely related to study drugs
Hypertension (Vascular disorders) | 0 (0) | 1 (2) — Grade 1, possibly related to study drugs
Hypertension (Vascular disorders) | 0 (0) | 1 (2) — Grade 1, possibly related to Ziv-Aflibercept
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Grade 2, possibly related to Ziv-Aflibercept
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) — Grade 1, unlikely related to study drugs
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Grade 2, possibly related to study drugs
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) — Grade 1, possibly related to study drugs
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 2, unlikely related to study drugs
Infusion related reaction (General disorders) | 1 (1) | 0 (0) — Grade 2, possibly related to study drugs
Infusion related reaction (General disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) — Grade 2, possibly related to study drugs
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3) — Grade 1, possibly related to study drugs
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) — Grade 1, possibly related to study drugs
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Platelet count decreased (Investigations) | 0 (0) | 2 (2) — Grade 1, possibly related to study drugs
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to Ziv-Aflibercept
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1, unlikely related to study drugs
Serum amylase increased (Investigations) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — Grade 2, unlikely related to study drugs
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Weight loss (Investigations) | 0 (0) | 1 (1) — Grade 1, possibly related to study drugs
Weight loss (Investigations) | 0 (0) | 1 (1) — Grade 1, unlikely related to study drugs
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 2, unlikely related to study drugs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02192541/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT02192541/Prot_SAP_001.pdf